CLINICAL TRIAL: NCT05747482
Title: Non-inferiority Randomized Clinical Trial Comparing Omenectomy and Omental Preservation in Resectable Gastric Cancer
Brief Title: Omentectomy vs Omental Preservation in Resectable Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Sandra Montmany-Vioque, MD, PhD, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMontmany2022
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cancer of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omentectomy (Other): Omentectomy during cancer gastric surgery
  Interventions: Other: Surgery procedure
- Omental preservation (Other): Preserval omentation during cancer gastric surgery
  Interventions: Other: Surgery procedure

INTERVENTIONS:
Other: Surgery procedure — Omentectomy vs omental preservations during gastric surgery
  Other Names: Omentectomy; Omental preservation

SUMMARY:
European clinical guidelines do not establish a clear recommendation neither for nor against omentectomy of this segment, the American clinical guidelines recommend omentectomy in view of its potential long-term oncological benefit, and Japanese clinical guidelines only recommend 2nd segment omentectomy in locally advanced gastric cancers (stage T3-T4) recommending omental preservation in early gastric cancers (stage T1-T2).

Faced with this lack of consensus, we propose a randomized, prospective and multicentric study in patients with resectable gastric cancer in stage T3-4 N+/- M0. Patients will be randomized into two groups, one where omentectomy of the 2nd omental portion will be performed and another where omental preservation will be performed.

The aim of our study is to analyze the disease-free interval and survival between both groups, also comparing postoperative complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Resectable gastric cancer
* Gastric cancer T3-4 N+/- M0

Exclusion Criteria:

* M1
* Non surgical patients for medical status
* Non resectable gastric cancer during surgery
* Endoscopic resectable gastric cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
disease free interval | 5 years
  time between surgery and recurrence. Units of measure: months

SECONDARY OUTCOMES:
global survival | 5 years
  survival between surgery and last follow-up date. Units of measure: percentage
survival at 5 years | 5 years
  survival between surgery and 5 years. Units of measure: percentage
complications - CCI | 30 days after surgery
  type of complications and CCI number. Units of measure: enter number between 1 and 100
postoperatory mortality | 30 days after surgery
  mortality after surgery. Units of measure: percentage

IPD SHARING:
Plan to Share IPD: Yes